CLINICAL TRIAL: NCT00594698
Title: A Familiarization and Safety Study of Myocardial Perfusion Contrast Echocardiography With PB127 Ultrasound Contrast Agent in Patients With Suspected Obstructive Coronary Artery Disease
Brief Title: Familiarization and Safety Study of PB127 Ultrasound Contrast Agent
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Point Biomedical (Industry)
Responsible Party: Tom Ottobonie, PhD/Chief Operating Officer, POINT Biomedical Corp.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127-005
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Disease
Keywords: Perfusion; Echocardiography; Cardiac angiography; SPECT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PB127 for injectable suspension — 0.175 mg/kg diluted in 150 mL 5% Dextrose for Injection in glass bottles, to be administered as a single continuous infusion during image acquisition. Infusion time not to exceed 60 minutes
  Other Names: CARDIOsphere®

SUMMARY:
The purpose of this study is to evaluate preparation and administration of PB127, echocardiographic images obtained during PB127 administration, and evaluate the safety of PB127.

DETAILED DESCRIPTION:
The primary objectives of this clinical trial are:

1. To train potential Phase 3 investigational sites in the preparation and andministration of PB127
2. To train potential Phase 3 investigational sites in the acquisition of adequate images
3. To collect additional safety information regarding intravenous administration of PB127
4. To obtain a larger sample of images obtained with the Acuson Sequoia ultrasound system.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Scheduled for stress echocardiography, SPECT nuclear imaging and/or coronary angiography within the two weeks prior to or following Study Day 1
3. Adequate visualization of all myocardial segments in at least one imaging plane during screening non-contrast echocardiogram

Exclusion Criteria:

1. Women who were pregnant or lactating
2. Known hypersensitivity or known contraindication to

   1. Dipyridamole
   2. Other ultrasound contrast agents
   3. Blood, blood products, albumin, egg, or protein
3. Use of caffeine or xanthine containing products within the 24 hours prior to PB127 MPE
4. Frequent (> 60/hour) or symptomatic ventricular ectopics at baseline
5. Atrial fibrillation
6. Permanent pacemaker or defibrillator
7. History of:

   1. Complex ventricular arrhythmia
   2. Chronic hepatitis
   3. Liver disease characterized by one or more of the following:

      * current jaundice
      * elevated bilirubin > upper limit of normal
      * currently elevated hepatic enzymes > 2X upper limit of normal
      * current or previous hepatic viral infection
   4. Chronic obstructive pulmonary disease (COPD) that, in the opinion of the Investigator, was significant enough to contraindicate dipyridamole
   5. Bronchospastic airway disease that, in the opinion of the Investigator, was significant enough to contraindicate dipyridamole
   6. Coronary artery bypass graft (CABG) within the 7 days prior to Study Day 1
   7. Heart transplant
   8. Q wave myocardial infarction within the 7 days prior to Study Day 1
   9. Cardiac intervention or surgery within the 7 days prior to Study Day 1
8. Hypertension (systolic blood pressure [SBP] >200 mmHg and diastolic blood pressure [DBP] >110 mmHg)
9. Hypotension (SBP <90 mmHg) documented within the 24 hours prior to Study Day 1
10. Significant valvular disease

    1. Severe aortic stenosis (>100 mmHg peak transvalvar gradient or <0.6 cm2 estimated valve area)
    2. Severe mitral regurgitation (usual clinical criteria plus or minus any of the following: proximal isovelocity surface area [PISA] >1 cm2, forward transmitral gradient of >2 m/sec, unexplained systolic flow reversal or blunting in the pulmonary veins)
    3. Severe mitral stenosis (<1.0 cm2 estimated valve area)
11. Congestive heart failure (New York Heart Association [NYHA] Class IV); NYHA classes are defined in Appendix D of the protocol (see Appendix 16.1.1)
12. Pulmonary edema within the 7 days prior to Study Day 1
13. Resting oxygen saturation of < 90%
14. Pulmonary hypertension characterized by estimated pulmonary artery systolic pressure of >50 mmHg by echo or catheter criteria on Study Day 1
15. Unstable angina, Canadian Cardiovascular Society (CCS) Class IV severity, with ongoing symptoms and/or ongoing infusion of intravenous nitroglycerin; CCS grading criteria are provided in Appendix E of the protocol (see Appendix 16.1.1)
16. Second degree heart block or greater
17. Use of intravenous or intracoronary contrast agent within the 24 hours prior to Study Day 1
18. Medical conditions or other circumstances that would significantly decrease the chances of obtaining reliable data or achieving the study objectives, ie, drug dependence, psychiatric disorder, dementia, or other reasons for expected poor compliance with the Investigator's instructions; medical conditions, associated illness, or extenuating circumstances that made it unlikely that a patient can complete the clinical trial or follow-up evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-02; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Technical adequacy and diagnostic quality of PB127 images | 24 hours

SECONDARY OUTCOMES:
Compliance with image acquisition and Pb127 administration procedures | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ehlgen, MD, PhD, Study Director — POINT Biomedical Corp.
Locations (34):
- United States (34):
  - Michael Morgan, MD, Phoenix, Arizona
  - Heartcare, P.C., Scottsdale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Long Beach VA Medical Center Cardiology Division, Long Beach, California
  - University of California San Diego Division of Cardiology, San Diego, California
  - San Francisco VA Medical Center NCIRE, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Washington Hospital Center Cardiovascular Research Institute, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - The Center for Cardiovascular Studies Kramer and Crouse Cardiology, Shawnee Mission, Kansas
  - Androscoggin Cardiovascular Associates, Auburn, Maine
  - Maine Cardiology Associates, South Portland, Maine
  - New England Medical Center, Boston, Massachusetts
  - Cardiovascular Consultants, Kansas City, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - MidWest Cardiologist Research, Columbus, Ohio
  - Endovascular Research, LLC, Eugene, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pittsburgh Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Austin Heart, Austin, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Methodist DeBakery Heart Center Cardiovascular Imaging Institute, Houston, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center Department of Cardiology, Seattle, Washington
  - Inland Cardiology, Spokane, Washington
  - Northwest Cardiovascular Research Institute Spokane Cardiology, Spokane, Washington